CLINICAL TRIAL: NCT02138487
Title: Restricted Convalescence: Outcomes Following Urogynecologic Procedures
Acronym: ReCOUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Kimberly Kenton, Professor of Obstetrics and Gynecology, Professor of Urology, Division Chief Female Pelvic Medicine and Reconstructive Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU00084995
Record Dates: First submitted 2014-05-08; First posted 2014-05-14 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; reconstructive pelvic surgery; postoperative restrictions; patient satisfaction
MeSH Terms: conditions — Pelvic Organ Prolapse; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restricted postoperative activity (Active Comparator): Women in the "restricted postoperative activity" group must abstain from exercise and heavy lifting for 3 months postoperatively
  Interventions: Other: Restricted postoperative activity
- Liberal postoperative activity (Experimental): Women in the "liberal postoperative activity" group will be allowed to resume their normal activities without restriction.
  Interventions: Other: liberal postoperative activity

INTERVENTIONS:
Other: liberal postoperative activity — Women will be given specific instructions regarding postoperative activities and will not have any limitations regarding activity.
  Arms: Liberal postoperative activity
Other: Restricted postoperative activity — Women in this group will be given instructions regarding postoperative activity and will need to abstain from heavy lifting, running, aerobics for 3 months.
  Arms: Restricted postoperative activity

SUMMARY:
The investigators are conducting a study to better understand the relationship between activity restrictions and women's satisfaction following urogynecologic surgery for prolapse. We hypothesize that women with less stringent postoperative restrictions will have higher levels of satisfaction 12 weeks following surgery with no difference in respect to anatomic outcome.

DETAILED DESCRIPTION:
Pelvic floor disorders (PFD) dramatically affect millions of women's quality of life (QOL), and 30% of American women will undergo reconstructive surgery for urinary incontinence or pelvic organ prolapse to improve bothersome symptoms and quality of life. Surgical goals of women with PFD is often to resume their normal activities, which they have limited secondary to bothersome symptoms. Yet, traditionally surgeons placed strict postoperative restrictions on patient's activity levels for 3 months; sometimes even recommending life long lifting and activity restrictions. Activity restrictions are imposed on the premise that exercise can "weaken" surgical healing; however, emerging data from other fields suggests that increased activity may actually promote the healing process. We aim to determine whether satisfaction, recovery, and anatomic outcomes after surgery are related to type of postoperative activity recommendations (liberal versus restricted). Women having surgery for PFD will be randomized to receive either liberal or restricted postoperative activity recommendations and satisfaction, symptoms, QOL and anatomic outcomes will be measured after surgery. We hypothesize that women with liberal activity recommendations will recover more quickly and report higher satisfaction and QOL, have fewer symptoms, and have similar anatomic outcomes to women with restricted activity restrictions. These data will change paradigms of women's health and recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory women undergoing surgical management of pelvic organ prolapse
* Prolapse > to Stage II on POP-Q
* Age >18 yrs
* Completed childbearing
* All subjects must have given signed, informed consent prior to registration on study
* All subjects must be able to read and complete study documents

Exclusion Criteria:

* Wheelchair-bound women
* Women with neurologic disease (Multiple Sclerosis, Parkinson's Disease)
* Abdominal approach with laparotomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-08; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction | 12 weeks following surgery
  Satisfaction will be assessed following reconstructive pelvic surgery for prolapse using a question which assesses a patient's global impression. Specifically, patients will be asked the question "how satisfied are you with your prolapse surgery?" at 12 wks to assess overall satisfaction. Possible responses include "completely satisfied," "mostly satisfied," "neutral," "mostly dissatisfied," and "completely dissatisfied."

SECONDARY OUTCOMES:
Anatomic Outcomes | 12 weeks and 1 year following surgery
  Anatomic outcomes will be assessed on physical examination 12 weeks and 1-year following reconstructive pelvic surgery.
Quality of Life | 12 weeks and 1 year following surgery
  Quality of life will be assessed using several validated questionnaires at 12 weeks and 1 year following reconstructive pelvic surgery for prolapse.
Pain | 12 weeks and 1 year following surgery
  Pain will be assessed using a visual analog scale at 12 weeks and 1 year following reconstructive pelvic surgery.
Activity level | 12 weeks and 1 year
  Activity level will be assessed using a validated questionnaire at 12 weeks and 1 year following reconstructive pelvic surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Kenton, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Virginia Tech Carilion School of Medicine, Roanoke, Virginia

REFERENCES:
- [Derived] Mueller MG, Collins SA, Lewicky-Gaupp C, Tavathia M, Kenton K. Restricted Convalescence Following Urogynecologic Procedures: 1-Year Outcomes From a Randomized Controlled Study. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):e336-e341. doi: 10.1097/SPV.0000000000000922. PMID 32947549
- [Derived] Bochenska K, Hall E, Griffith JW, Kenton K, Alverdy A, Lewicky-Gaupp C, Mueller M. The Promise of PROMIS in Pelvic Organ Prolapse. Female Pelvic Med Reconstr Surg. 2019 Nov-Dec;25(6):426-429. doi: 10.1097/SPV.0000000000000685. PMID 30570502
- [Derived] Mueller MG, Lewicky-Gaupp C, Collins SA, Abernethy MG, Alverdy A, Kenton K. Activity Restriction Recommendations and Outcomes After Reconstructive Pelvic Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2017 Apr;129(4):608-614. doi: 10.1097/AOG.0000000000001924. PMID 28277355